CLINICAL TRIAL: NCT06372795
Title: Effect of Early Progressive Resistance Swallowing Training on Swallowing Related Muscle Strength in Patients With Tracheotomy
Brief Title: Resistance Swallowing Training in Patients With Tracheotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KY2023635
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Swallowing Training on Muscle Strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Other: pure effortful swallowing
- Test group (Experimental)
  Interventions: Other: progressive resistance swallowing training

INTERVENTIONS:
Other: pure effortful swallowing — The investigator instructed the patient to "swallow forcefully while squeezing the tongue upward and backward in the direction of the soft palate" based on the sounds of an electronic timer.
  Arms: Control group
Other: progressive resistance swallowing training — Patients in the test group, resistance swallowing exercise was performed by providing external resistance through Iowa Oral Performance Instrument (IOPI), and all other protocols were performed the same as those in the control group.
  Arms: Test group

SUMMARY:
The goal of this clinical trial is to learn investigate the effect of instrument-assisted early progressive resistance swallowing training on swallowing related muscle strength in critically ill patients. It will also learn about the safety of swallowing training. The main questions it aims to answer are:

* Does instrument-assisted early progressive resistance swallowing training increase the swallowing related muscle strength in critically ill patients?
* What medical problems do participants have when taking swallowing training?

Researchers will compare instrument-assisted early progressive resistance swallowing training to pure effortful swallowing to see if instrument-assisted early progressive resistance swallowing training works to increase muscle strength.

Participants will:

-Take instrument-assisted early progressive resistance swallowing training or pure effortful swallowing every day for 2 weeks and take muscle strength test every week.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Tracheotomy after intubation and ventilator ventilation
* Receiving treatment in ICU, and expected hospital stay > 2 weeks after pneumonectomy
* Be able to cooperate to complete the maximum anterior tongue pressure test

Exclusion Criteria:

* Inability to cooperate with tongue pressure testing and swallowing training, including disturbance of consciousness, oropharyngeal neuromuscular or motor impairment
* Patients refuse to participate in this study
* Significant malocclusion and facial asymmetry

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Forced swallowing tongue pressure | Day 14 after training
  Place the pressure balloon on the prelingual pressure measurement site. The examiner placed the water in the participant 's mouth using a disposable 3 mL syringe. Subjects held 3 mL of water in their mouth and swallowed as forcefully as possible as directed by the examiner to observe instrument readings.

IPD SHARING:
Plan to Share IPD: No